CLINICAL TRIAL: NCT06399328
Title: Cardiovascular Risk Stratification on the Basis of Surface Enhanced Raman Spectroscopy. Assessment of Technology for Early Subclinical Detection of Coronary Heart Disease Based on Serum Metabolic Shifts .
Brief Title: Cardiovascular Risk Stratification on the Basis of Surface Enhanced Raman Spectroscopy
Acronym: CRUISERS
Status: Recruiting | Type: Observational
Sponsor: Samara State Medical University (Other)
Collaborators: Samara Regional Clinical Hospital V.D. Seredavin (Other)
Responsible Party: Sponsor
Other Study IDs: ATSERS001
Record Dates: First submitted 2024-04-18; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Coronary Atherosclerosis of Native Coronary Artery
Keywords: Surface Enhances Raman Spectroscopy; Computer Tomography of coronary arteries; Calcium coronary score; cardiovascular risk stratification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Serum samples 2 ml of each person for SERS evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A group (normal coronary arteries): A group: no signs of coronary calcium (<75 percentile values of corresponding age and gender ) and no plaques (normal coronary arteries)
  Interventions: Diagnostic Test: Surface Enhanced Raman Spectroscopy
- B group (subclinical coronary atherosclerosis, stage 1): B group: coronary calcium >75 percentile of corresponding age and gender /or plaques on MSCT without stenosis
  Interventions: Diagnostic Test: Surface Enhanced Raman Spectroscopy
- C group ( subclinical/clinically evident coronary atherosclerosis,stage 2): C group: atherosclerotic plaques of coronary artery with stenosis 50% and more, with or without chest pain
  Interventions: Diagnostic Test: Surface Enhanced Raman Spectroscopy

INTERVENTIONS:
Diagnostic Test: Surface Enhanced Raman Spectroscopy — Spectral measurements of blood serum were performed on a silver nanoparticle substrate. Serum samples were collected and placed in sterile tubes with subsequent freezing at -18°C. Immediately before analysis, samples were thawed at room temperature. For spectral analysis, each 1.5 μL serum sample was applied to a substrate with a layer of silver nanoparticles and dried for 30 minutes. The spectral characteristics of serum were analyzed using an experimental bench consisting of a spectrometric system and a microscope (ADF U300, ADF, China). The spectra were excited in the near infrared range using a laser module with a center wavelength of 785 nm. Each of the obtained spectra represented a discrete set of 1700 parameters in the range of studied frequencies.

SUMMARY:
In the modern population, mortality and disability from cardiovascular diseases is predominant and is realized as a major medical and social problem. The study of mechanisms of development of age-related diseases, such as coronary heart disease (CHD), has demonstrated multiple qualitative and quantitative changes of metabolites in biological fluids of the body - blood, in the vascular wall, as well as in the tissues of vital organs. In routine clinical practice only about a dozen metabolic parameters are determined by standard laboratory methods.

The proposed approach belongs to a new scientific direction , wich development is aimed at individualization of approaches to risk stratification of cardiovascular diseases and their complications. The data obtained in this project will allow to create a base of medical knowledge about spectral characteristics of blood serum, which most fully reflect the metabolic profile associated with atherosclerosis of coronary arteries. Researchers offer so-called multiplex diagnostics when multiple parameters of a biological object obtained by serum biochemical analysis and optical scattering analysis are used. Recognition of this big data is possible only by methods of mathematical analysis, which can take into account the degree of deviations, their directionality in each point of the spectral characteristic.

Until recently, the standard setup for Raman light scattering studies had significant dimensions. The high cost of such installations made it difficult to widely use the method of optical spectroscopy for rapid analysis of medical objects. In recent years, the situation on the market of scientific instrumentation has changed radically, which allowed to significantly reduce and cheapen all components of Raman installations.This simplification and cheapening allows to bring optical research in medicine (optical biopsy) to a new level of use, directly into clinical laboratories.

Novelty: This area of research belongs to high-tech and is very little represented in Europe. The prospect of using Surface Enhanced Raman spectroscopy (SERS) to determine subclinical lesions of coronary arteries and for risk stratification of diseases associated with atherosclerosis is quite unique and wasn't explored yet.

DETAILED DESCRIPTION:
Currently, multispiral computed tomography of coronary arteries (MSCT) is the most informative method for diagnosing subclinical CHD, as well as in symptomatic patients (gold standard method). Investigators are interested in including all patients who have undergone coronary artery MSCT within the last year, who will be divided into groups:

1. Those with no cardiac pain at baseline and the diagnosis of CHD was not established before MSCT and was not confirmed by the MSCT result. Patients without any pain syndrome.
2. Those with initial cardiac pain considered as atypical angina pectoris but IBS not confirmed by MSCT.
3. Those in whom the initial cardiac pain was considered as atypical angina and the diagnosis of CHD was confirmed by MSCT.
4. Those in whom the diagnosis of CHD was verified before MSCT and confirmed by MSCT.

According to the results of MSCT, all included will be divided into a group without CHD and two groups with CHD:

1. - without clinical manifestations of CHD with low calcium score and without plaques (without signs of CHD)
2. - without clinical manifestations of CHD with high calcium count, presence of plaques and without stenosis (subclinical CHD)
3. -with clinical manifestations of CHD with high calcium count, plaques and stenoses of different degrees (clinical CHD).

Accordingly, the differences of Raman spectrum in these groups will be revealed, which will make it possible to determine the degree of coronary atherosclerosis severity and stratify cardiovascular risk with a certain accuracy based only on the blood serum spectrum. These data will undoubtedly be of high scientific and practical value. To our knowledge, no similar studies have been conducted in the world.

No additional invasive procedures are anticipated in this study. A single blood draw is performed from the catheter before contrast injection for MSCT using a certified technique.

Aim: To propose a technology for early diagnosis of CHD and cardiovascular risk stratification based on serum metabolic shifts determined by serum Raman spectroscopy.

Objectives:

1. To study the features of Surface Enhanced Raman spectrum ( SERS) depending on belonging to 1)group without CHD; 2)group with subclinical CHD; 3)group with CHD.
2. To determine the possibility of reliable division of patients into these groups using the model based on SERS and SERS model in combination with known clinical parameters using artificial intelligence methodology.
3. To propose a model of CHD risk stratification based on the obtained data.

ELIGIBILITY:
Inclusion Criteria:men and women who underwent MSCT of coronary arteries (CA) within the last year with determination of Agatston index and coronary plaques/ stenoses from 30 to 65 years old without verified diagnosis of coronary heart disease. (220 patients).

* without cardiac pain
* with atypical angina pectoris.
* with typical angina pectoris .
* possibly with asymptomatic atherosclerosis of carotid and other peripheral arteries not subject to surgical treatment (degree of stenosis not more than 50%) Possible combination with known type 2 diabetes mellitus not requiring insulin therapy, with hypertension stages 1-2.

Exclusion Criteria:-absence of MSCT CA results; poor image quality.

* tachycardia, irregular heart rhythm
* known at the time of inclusion: Acute Coronary Syndrom, myocardial infarction,any form of verified CHD, operated for coronary atherosclerosis (PCI) peripheral arteries (carotid, renal, leg),stroke of any kind.
* established diagnosis or clinical signs of chronic heart failure.
* familial hypercholesterolemia (total cholesterol 7.5 mmol/L or more),
* Type 1 diabetes mellitus (DM) or type 2 DM requiring insulin therapy
* Creatinine 135 µmol/L or higher;
* oncologic diseases, cirrhosis ,
* obesity : body mass index (BMI) 35kg/m2 and above,
* anemia Hemoglobin below 110g/l,
* dementia disorders,
* absence of informed consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators plan to include all patients who were clinically evaluated and underwent coronary artery MSCT within the last year, divided into groups:
  1. Those with no cardiac pain at baseline and the diagnosis of CHD was not established before MSCT and was not confirmed by the MSCT result. Patients without any pain syndrome.
  2. Those with initial cardiac pain considered as atypical angina pectoris but CHD not confirmed by MSCT.
  3. Those in whom the initial cardiac pain was considered as atypical angina and the diagnosis of CHD was confirmed by MSCT.
  According to the results of MSCT CA, all included will be divided into a group without CHD (A group) and two groups with CHD(B and C groups)
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Model for determination of normal (A) coronary anatomy, subclinical stage 1 (B)of atherosclerosis and stage 2 lesions on the base of surface enhanced Raman spectroscopy | 1 year
  Sensitivity and specificity will be calculated for models, discriminating status of coronary arteries on the basis of SERS. In a case of high model performance it would be possible to assess coronary lesions by serum samples only.

CONTACTS AND LOCATIONS:
Overall Officials: Petr A Lebedev, professor, Principal Investigator — chief of therapy chair of professional education department
Locations (1):
- Regional Samara clinical hospital na V.D.Seredavin, Samara, Samara Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Khristoforova YA, Bratchenko LA, Skuratova MA, Lebedeva EA, Lebedev PA, Bratchenko IA. Raman spectroscopy in chronic heart failure diagnosis based on human skin analysis. J Biophotonics. 2023 Jul;16(7):e202300016. doi: 10.1002/jbio.202300016. — https://pubmed.ncbi.nlm.nih.gov/36999197/
- See also: Bratchenko LA, Bratchenko IA, Khristoforova YA, Artemyev DN, Konovalova DY, Lebedev PA, Zakharov VP. Raman spectroscopy of human skin for kidney failure detection. J Biophotonics. 2021 Feb;14(2):e202000360. doi: 10.1002/jbio.202000360. — https://pubmed.ncbi.nlm.nih.gov/33131189/